CLINICAL TRIAL: NCT03535818
Title: Adjunctive GP Ablation In Redo-PVI: Paroxysmal Atrial Arrhythmias After Pulmonary Vein Isolation Are Driven By Ectopy-Triggering Left Atrial Ganglionated Plexus
Brief Title: Adjunctive Ganglionated Plexus Ablation in Redo-Pulmonary Vein Isolation
Acronym: ADD-GP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17HH3712
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Paroxysmal Atrial Fibrillation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, prospective study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Redo pulmonary vein isolation (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation
- Ganglionated plexus ablation + redo pulmonary vein isolation (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — RF application to achieve complete pulmonary vein isolation +/- ganglionated plexus ablation

SUMMARY:
The investigator propose to test the efficacy of adjunctive ET-GP ablation in patients undergoing redo PVI for paroxysmal AF.

DETAILED DESCRIPTION:
Patients with ongoing paroxysmal arrhythmias after pulmonary vein isolation (PVI) for paroxysmal and persistent atrial fibrillation (AF) get incrementally less benefit with redo-PVI. This implies non-pulmonary vein (PV) triggers, which are more challenging to locate. The autonomic nervous system is implicated in the multifactorial pathogenesis of AF but few studies have attempted neural targeting as a therapeutic intervention. We have demonstrated that stimulation of specific left atrial ganglionated plexi (GPs) triggers both AF and atrial ectopy and importantly stimulation of these sites may not induce AV block, the 'conventional' marker used to locate GPs. Having shown that these ectopy-triggering GP (ET-GP) sites are anatomically stable and can be rendered inactive by either ablation at the site or by ablation between the site and the adjacent PV, a single centre study suggests that ET-GP ablation can prevent recurrent AF in some patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females eighteen (18) to eighty five (85) years old
* Paroxysmal atrial fibrillation
* Previous pulmonary vein isolation
* Suitable candidate for catheter ablation
* Signed informed consent

Exclusion Criteria:

* Contraindication to catheter ablation
* Presence of a cardiac thrombus
* Valvular disease that is grade moderate or greater
* Any form of cardiomyopathy
* On amiodarone therapy
* Patients who lack capacity
* Active gastrointestinal bleeding
* Active infection or fever
* Renal failure (Creatinine >200µmol/L)
* Life expectancy shorter than the duration of the trial
* Bleeding or clotting disorders or inability to receive heparin
* Pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Any atrial arrhythmia >30s documented on ECGs | 12 months
  After blanking period 3 months

SECONDARY OUTCOMES:
Symptom recurrence requiring repeat ablations | 12 months
Complications | 12 months
Radiofrequency time | Within ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, PhD, Principal Investigator — Imperial College London
Locations (1):
- Prapa Kanagaratnam, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No